CLINICAL TRIAL: NCT02324816
Title: Non-Invasive Fat Layer Reduction in the Lateral Thighs With a Cryolipolysis System Using a Colder Treatment Parameter
Brief Title: Fat Layer Reduction in the Lateral Thighs Using CoolSculpting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeltiq Aesthetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZA14-005
Record Dates: First submitted 2014-12-05; First posted 2014-12-24 (Estimated); Results first posted 2020-09-24 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2020-09

CONDITIONS: Body Fat Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Lateral Thigh Treatment Group (Experimental): CoolSculpting treatment in the lateral thighs for non-invasive subcutaneous fat reduction.
  Interventions: Device: The Zeltiq CoolSculpting System

INTERVENTIONS:
Device: The Zeltiq CoolSculpting System — The CoolSculpting System delivers non-invasive cooling for the reduction of subcutaneous fat.

SUMMARY:
Evaluate the performance of a cryolipolysis system using a colder treatment parameter for non-invasive reduction of subcutaneous fat in the lateral thighs.

DETAILED DESCRIPTION:
Evaluation of the Zeltiq CoolSculpting System for non-invasive subcutaneous fat reduction in the lateral thighs.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects > 22 years of age and < 65 years of age.
* Subject has clearly visible fat on the intended treatment area (lateral thighs), which in the investigator's opinion, may benefit from the treatment.
* Subject has not had weight change exceeding 10 pounds in the preceding month.
* Subject with body mass index (BMI) up to 35. BMI is defined as weight in pounds multiplied by 703 divided by the square of the height in inches.
* Subject agrees to maintain his/her weight (i.e., within 5%) by not making any major changes in their diet or exercise routine during the course of the study.
* Subject has read and signed a written informed consent form.

Exclusion Criteria:

* Subject has had a surgical procedure(s) in the area of intended treatment.
* Subject has had an invasive fat reduction procedure (e.g., liposuction, mesotherapy) in the area of intended treatment.
* Subject has had a non-invasive fat reduction and/or body contouring procedure in the area of intended treatment within the past 4 months.
* Subject needs to administer, or has a known history of subcutaneous injections into the area of intended treatment (e.g., heparin, insulin) within the past month.
* Subject has a known history of cryoglobulinemia, cold urticaria, or paroxysmal cold hemoglobinuria.
* Subject has a known history of Raynaud's disease, or any known condition with a response to cold exposure that limits blood flow to the skin.
* Subject has a history of bleeding disorder or is taking any medication that in the investigator's opinion may increase the subject's risk of bruising.
* Subject is taking or has taken diet pills or supplements within the past month.
* Subject has any dermatological conditions, such as moderate to excessive skin laxity, or scars in the location of the treatment sites that may interfere with the treatment or evaluation (stretch marks is not an exclusion).
* Subject has an active implanted device such as a pacemaker, defibrillator, or drug delivery system
* Subject is pregnant or intending to become pregnant during the study period (in the next 4 months).
* Subject is lactating or has been lactating in the past 6 months.
* Subject is unable or unwilling to comply with the study requirements.
* Subject is currently enrolled in a clinical study of any other unapproved investigational drug or device.
* Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-11-14 (Actual); Primary Completion 2015-03-13 (Actual); Study Completion 2015-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Bachelor, MD, Principal Investigator — Innovation Research Center
Locations (1):
- Innovation Research Center, Pleasanton, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Lateral Thigh Treatment Group: Non-invasive subcutaneous fat reduction in the lateral thighs treatment group
  The Zeltiq CoolSculpting System: CoolSculpting treatment.
Period: Overall Study
Arm/Group | Lateral Thigh Treatment Group
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Female subjects with visible fat bulges on the outer thighs were recruited for the study.
Groups:
- Lateral Thigh Treatment Group: Non-invasive subcutaneous fat reduction in the lateral thighs treatment group using the CoolSculpting System.
Arm/Group | Lateral Thigh Treatment Group
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 45.0 [31 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 0
  Asian | 2
  Caucasian | 16
  Hispanic | 0
  Others | 1
Region of Enrollment [Number; unit: participants]
  United States | 19
Body Mass Index [Mean (Full Range); unit: kg//m^2^] | 26.5 [21 to 32.1]

OUTCOME MEASURES:

1. Primary Outcome: Safety of the Zeltiq CoolSculpting System in the Outer Thighs
Description: Tabulation of device and/or procedure-related adverse events and unanticipated adverse device effects will be performed. Adverse event information will be collected from the time of study enrollment through the 12 week follow-up visit. The Investigator will determine if an adverse event is related to the device and/or study procedure.
Time Frame: Enrollment through 12 week post-final treatment follow-up visit
Measure: Number; unit: events
Arm/Group | Lateral Thigh Treatment Group
Number analyzed (Participants) | 19
events
  Device and/or procedure related AEs | 8
  UADEs reported | 0

2. Secondary Outcome: Percentage of Correctly Identified Pre-treatment Photographs
Description: Change in the treated vs. untreated areas will be assessed by observation of changes in surface contour and/or fat volume by an independent photo review of pre-treatment and post-treatment images of the treated areas. Reviewers will be practicing dermatologists or plastic surgeons. All reviewers will be blinded to post-treatment vs. baseline untreated area. The order in which images will be presented will be randomized; for each subject placement of the baseline, pre-treatment image will be randomized for each pair of subject images. Reviewers will be asked to select the baseline photos for each subject photo series and record selections on a data collection form. Success is defined as at least 70% correct identification of pre-treatment images by 2 out of 3 reviewers.
Time Frame: 12 weeks post-final treatment
Population: Photo pairs for 19 subjects were reviewed by blinded reviewers.
Measure: Count of Units; unit: photo pairs
Units Other Than Participants: photo pairs
Arm/Group | Lateral Thigh Treatment Group
Number analyzed (Participants) | 19
Number analyzed (photo pairs) | 19
photo pairs | 14
Statistical Analysis 1: Comparison: Lateral Thigh Treatment Group; Test type: Other; success proportion = 73.7, 95% CI 2-sided [48.8 to 90.9]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from enrollment through the 12-week post-treatment follow-up visit.
Description: An adverse event is defined as any untoward medical occurrence in a subject, regardless of whether the event is related to the device or the treatment.
Arm/Group | Lateral Thigh Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 14/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lateral Thigh Treatment Group (N=19)
Prolonged swelling (Skin and subcutaneous tissue disorders) | 4 (4) — Prolonged swelling in the treatment area that had a duration of >1 month.
Prolonged bruising (Skin and subcutaneous tissue disorders) | 2 (2) — Bruising on the outer thigh that persisted >1 month.
Erythema lasting > 2 weeks (Skin and subcutaneous tissue disorders) | 2 (2) — Erythema in the treatment are that persisted > 2 weeks.
Cold with cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Cold with cough reported. Duration approximately 1 week.
24 hour cold (General disorders) | 1 (1) — Head cold of 24 hour duration
Rotator cuff pin adjustment (Surgical and medical procedures) | 1 (1) — Rotator cuff pin adjusted
Tendonitis flare up (Musculoskeletal and connective tissue disorders) | 1 (1) — Tendonitis in left wrist reportedly flared during study period.
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) — Eczema reported on left hand.
Menopausal changes (Reproductive system and breast disorders) | 1 (1) — Menopausal symptoms of fatigue reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No